CLINICAL TRIAL: NCT03494387
Title: Hyperoxia and Antioxidants During Major Non-cardiac Surgery and Risk of Cardiovascular Complications, a Blinded 2x2 Factorial Randomised Clinical Trial
Brief Title: VitamIn and oXygen Interventions and Cardiovascular Events
Acronym: VIXIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Cecilie Petersen, MD, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: VIXIE2018
Record Dates: First submitted 2018-03-21; First posted 2018-04-11 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Cardiac Complication
Keywords: Antioxidant; Hyperoxia; Troponin; MINS; Ascorbic acid; N-acetylcysteine
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen; Antioxidants; Ascorbic Acid; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Oxygen; Drug: Antioxidants
- 2 (Experimental)
  Interventions: Drug: Oxygen; Drug: Antioxidants

INTERVENTIONS:
Drug: Oxygen — 80% versus 30% inspiratory oxygen concentration
Drug: Antioxidants — Antioxidants versus placebo
  Other Names: Ascorbic acid; N-acetylcysteine

SUMMARY:
This study examines the risks and benefits of antioxidants and normal versus high inspiratory oxygen fraction during anaesthesia.

DETAILED DESCRIPTION:
Adult patients with risk factors for developing postoperative cardiac complications will be enrolled in the study. The patients will be randomised to receiving antioxidants or placebo perioperatively and 30% or 80% inspiratory oxygen concentration during anaesthesia and 2 hours postoperatively. The primary outcome is MINS (myocardial injury after non-cardiac surgery). The antioxidants are ascorbic acid (vitamin C) 3 grams intravenously preoperatively and N-acetylcysteine 100 milligrams/kilogram body weight intravenous infusion for 4 hours, starting at the same time as anaesthesia.

The study is a long-term follow-up study of the risk of mortality, MI and readmissions performed at 1 year after inclusion of the last patient. Two other follow-up studies are planned: One investigation of ischaemic troponin elevations defined as peak troponin levels above the internationally defined thresholds without extracardiac causes; another investigating the intervention effects in the subgroup of patients undergoing vascular surgery with specific emphasis on episodes of intraoperative hypotension within the following thresholds: MAP below 70 mmHg, 65 mmHg, 60 mmHg and 55 mmHg.

ELIGIBILITY:
Inclusion criteria:

All of the listed criteria (1.-4.) must be met.

1. Age 45 years or above
2. Elective or acute surgery in general anaesthesia
3. Scheduled for abdominal, orthopaedic, or vascular surgery with expected surgery duration of one hour or more.
4. Fulfil any 1 of the following 5 criteria:

   1. - History of coronary artery disease including angina
   2. - History of stroke
   3. - Undergoing vascular surgery
   4. - History of peripheral arterial disease
   5. - Any 2 of the following 8 criteria: i. Acute surgery ii. Current or previous daily smoking iii. History of hypertension iv. Diabetes mellitus requiring medical treatment v. History of transient cerebral ischemia vi. Plasma creatinine >175 µM vii. Age 70 years or above viii. History of congestive heart failure

Exclusion criteria:

1. Surgery within 30 days prior to operation
2. Arterial oxygen saturation below 90% without oxygen supplementation
3. Inability to give informed consent
4. Drug allergy towards any of the drugs involved in the trial
5. Previous treatment with bleomycin
6. Pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Myocardial injury after non-cardiac surgery (MINS) | 30 days
  Troponin measurement the first 3 postoperative days. Assessed by area under the curve.

SECONDARY OUTCOMES:
Mortality | During the study period until completion of last visit of last patient
  Assessed as time to event analysis
Non-fatal myocardial infarction | During the study period until completion of last visit of last patient
  Assessed as time to event analysis
Non-fatal Serious Adverse Event | During the study period until completion of last visit of last patient
  Assessed as time to event analysis

OTHER OUTCOMES:
Surgical site infection | Assessed at postoperative day 30
  Infection in surgical area as defined by the Center for Disease Control
Pneumonia | Assessed at postoperative day 30
  Pneumonia as defined by the Center for Disease Control
Sepsis | Assessed at postoperative day 30
  Sepsis as defined by the joint task force by the European Society of Intensive Care Medicine and the Society of Critical Care Medicine
Acute respiratory failure | Assessed at postoperative day 30
  Acute respiratory failure defined as the need for controlled ventilation or oxygen saturation of 900% or less despite of oxygen therapy
Acute kidney injury | Assessed at postoperative day 30
  Acute kidney injury as defined Kidney Disease Improving Global Outcomes guidelines

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Abdominalcentret, Rigshospitalet, Copenhagen
  - HovedOrtoCentret, Rigshospitalet, Copenhagen
  - Bispebjerg and Frederiksberg Hospital, University of Copenhagen, Copenhagen
  - Herlev Hospital, Herlev

REFERENCES:
- [Derived] Loft FC, Holse C, Aasvang EK, Vester-Andersen M, Rasmussen LS, Jorgensen LN, Meyhoff CS. Effects of Hyperoxia and Antioxidants on Mortality, Hospital Admissions, and Myocardial Infarction After Noncardiac Surgery: 1-Year Follow-Up of a Randomized Controlled Trial. Acta Anaesthesiol Scand. 2025 Nov;69(10):e70118. doi: 10.1111/aas.70118. PMID 41055553